CLINICAL TRIAL: NCT01219218
Title: Shockwave Treatment for Advanced Angina in Maastricht (SWAAM). A Pilot Study
Brief Title: Extracorporeal Shockwave Therapy for the Treatment of Advanced Angina Pectoris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medispec (Industry)
Collaborators: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESMR-AZM-NL
Record Dates: First submitted 2010-10-10; First posted 2010-10-13 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Refractory Angina Pectoris
Keywords: Extracorporeal Shockwave Therapy; Myocardial Ischemia; Refractory Angina
MeSH Terms: conditions — Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Treatment group. Patients in this group receive actual shockwave therapy.
  Interventions: Device: Cardiac Extracorporeal Shockwave Therapy generator (Cardiospec)

INTERVENTIONS:
Device: Cardiac Extracorporeal Shockwave Therapy generator (Cardiospec) — Energy Density - 0.09 mJ/mm2
  Other Names: Cardiospec; ESMR therapy; Extracorporeal Shockwave Myocardial Revascularization

SUMMARY:
Low intensity shockwaves have been proven in animal studies to induce local growth of new blood vessels from existing ones.

The hypothesis of this study is that shockwave therapy could improve the symptoms of patients with refractory angina not amenable to revascularization with angioplasty or bypass surgery.

DETAILED DESCRIPTION:
Low intensity shockwaves (1/10 the ones used in Lithotripsy) are delivered to myocardial ischemic tissue. Shockwaves are created by a special generator and are focused using a shockwave applicator device. The treatment is guided by standard echocardiography equipment. The shockwaves are delivered in synchronization with Patient R-wave to avoid arrhythmias. The treatment is painless.

At first, the patient undergoes stress-SPECT testing to identify the ischemic areas. Following that, the same area is localized by the ultra-sound device and the shockwaves are focused to the ischemic area. Several treatment session (9 in total, spread over 9 weeks) are required for optimal results.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with chronic stable angina pectoris, for a period of at least 3 months. Diagnosis is based on medical history, complete physical evaluation.
* Patient has documented myocardial segments with reversible ischemia.
* Patient is classified in AP CCS of III-IV.
* Patient should be on a stable dosage of medication used to treat angina for at least 6 weeks prior to enrollment.
* Patient demonstrates exercise tolerance capacity of no higher than 125 W on a modified Bruce treadmill exercise test until presence of clinical symptoms (i.e. angina, ST-depression).
* Patient demonstrates exercise tolerance time and stability averaging no more than 25% of each other (the tests will be performed within two weeks and at least a day different between the two).
* Patient has documented epicardial coronary artery disease not amenable to angioplasty or CABG.
* Patient has signed an IRB approved informed consent form.
* Patient's condition should be stable and should have a life expectancy of >12 months. Patient's current and past medical condition and status will be assessed using previous medical history, physical evaluation, and the physicians (principle investigator's) medical opinion.

Exclusion Criteria:

* Patient is pregnant
* Patient has chronic lung disease including emphysema and pulmonary fibrosis.
* Patient has active endocarditis, myocarditis or pericarditis.
* Patient is simultaneously participating in another device or drug study, or has participated in any clinical trial involving an experimental device or drug, including other drugs or devices enhancing cardiac neovascularization, or any ESWT machine of a competitor company within 3 months of entry into the study.
* Patients who are unwilling or unable to cooperate with study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Time to Angina | 6 months
  Change in time to angina using the modified Bruce exercise test from baseline to the 6 months post baseline assessment

SECONDARY OUTCOMES:
Change in SPECT | 6 months
  The change in perfusion in pharmacological induced stress SPECT test (at rest and at stress) from baseline to 6 months post baseline (17 segment model)
Change in AP-CCS | 6 months
  The AP-CCS stage at the 6 months post baseline.
Total Exercise time | 6 months
  The change in total exercise time (Exercise Tolerance Test- ETT) from baseline to 6 months post baseline.
Number of Angina attacks (patient diary) | 6 months
  The change in the number of angina attacks from baseline to 6 months post baseline. The number of attacks per week will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Johannes Waltenberger, MD, PhD, Principal Investigator — Academisch Ziekenhuis Maastricht
Locations (1):
- Academisch Ziekenhuis Maastricht, Maastricht, Netherlands